CLINICAL TRIAL: NCT01181297
Title: Double Blind Controlled Trial of an Extensively Hydrolyzed Formula With a Probiotic vs. an Extensively Hydrolyzed Formula Without a Probiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Other Study IDs: 3369-2
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Allergy
Keywords: Confirmed milk allergy
MeSH Terms: conditions — Hypersensitivity

ARMS (2):
- Extensively Hydrolyzed Formula with a Probiotic (Experimental): Extensively Hydrolyzed Formula with a Probiotic
  Interventions: Other: Extensively Hydrolyzed Formula with a Probiotic
- Extensively Hydrolyzed Formula without a Probiotic (Placebo Comparator)
  Interventions: Other: Extensively Hydrolyzed Formula without a Probiotic

INTERVENTIONS:
Other: Extensively Hydrolyzed Formula with a Probiotic
  Arms: Extensively Hydrolyzed Formula with a Probiotic
Other: Extensively Hydrolyzed Formula without a Probiotic
  Arms: Extensively Hydrolyzed Formula without a Probiotic

SUMMARY:
The purpose of this study is to confirm the hypoallergenicity of an extensively hydrolyzed formula with an added probiotic in children with documented milk allergy.

ELIGIBILITY:
Inclusion Criteria:

* ≤14 years of age
* Essentially asymptomatic for a minimum of 7 days pre-challenge.
* Successful previous consumption of Extensively Hydrolyzed Formula within 1 week of study enrollment
* Medically documented allergy to cow's milk

Exclusion Criteria:

* Presence of underlying systemic disease or other illness
* Used Beta-blockers within 12-24 hours of challenges
* Use of short-acting antihistamines within 3 days
* Use of medium-acting antihistamines within 7 days
* Use of long-acting antihistamines within 6 weeks
* Use of oral steroid medication within 3 weeks

Max Age: 14 Years
Age Groups: Child
Dates: Start 2003-01; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Dept. of Paediatrics, Azienda Ospedaliera di Padova, Padua, Veneto, Italy
- Wilhelmina Children's Hospital, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Muraro A, Hoekstra MO, Meijer Y, Lifschitz C, Wampler JL, Harris C, Scalabrin DM. Extensively hydrolysed casein formula supplemented with Lactobacillus rhamnosus GG maintains hypoallergenic status: randomised double-blind, placebo-controlled crossover trial. BMJ Open. 2012 Mar 5;2(2):e000637. doi: 10.1136/bmjopen-2011-000637. Print 2012. PMID 22396223